CLINICAL TRIAL: NCT01714648
Title: An Uncontrolled, Open-label Feasibility Study to Demonstrate That a GnRH Agonist (Decapeptyl) Can be Safely Administered to Trigger Final Oocyte Maturation in High Responder Patients to Mitigate the Risk of OHSS
Brief Title: Can GnRH Agonist Trigger Prevent Ovarian Hyperstimulation Syndrome?
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated: recruiting or enrolling participants has halted prematurely and will not resume; participants are no longer being examined or treated
Sponsor: Elisha Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Dr. Shahar Kol, Principal Investigator, Elisha Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MSD-ELISHA1; 8328-086 (Other Grant/Funding Number: MSD Database number 50036)
Record Dates: First submitted 2012-10-20; First posted 2012-10-26 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Ovarian Hyperstimulation Syndrome
Keywords: OVULATION INDUCTION
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OHSS high risk patients (Experimental): Triptorelin 0.2 mg
  Interventions: Drug: Triptorelin 0.2 mg

INTERVENTIONS:
Drug: Triptorelin 0.2 mg — A single bolus of 0.2 mg triptorelin given 34-36 hours before oocyte retrieval.
  Other Names: Decapeptyl 0.2 mg

SUMMARY:
Ovarian hyperstimulation syndrome (OHSS) is a major complication of ovarian stimulation for IVF if hCG is used to trigger final oocyte maturation. The investigators propose that using GnRH agonist as a trigger will eliminate OHSS, even in high-risk patients.

DETAILED DESCRIPTION:
Administration of hCG (10.000 or 5.000 IU) is essential in IVF protocols to trigger final oocyte maturation after ovarian stimulation. In high responder patients with potential risk of developing OHSS, hCG is usually withheld and the treatment cycle is cancelled without obtaining (cryopreserved) embryos for replacement.

An alternative approach to trigger final oocyte maturation is to administer a GnRH agonist instead of hCG. This method is not possible following a long GnRH agonist protocol which causes down-regulation of the GnRH receptor. However, following GnRH antagonist treatment the GnRH receptor remains receptive to competitive binding by a GnRH agonist.

It has been well-described in earlier IVF trials that a bolus of GnRH agonist will displace the GnRH antagonist from the GnRH receptors in the pituitary inducing an endogenous LH (and FSH) surge resulting in the maturation of oocytes and good quality embryos. In addition, the risk of moderate-to-severe ovarian hyperstimulation syndrome (OHSS) becomes minimal due to the rapid demise of the corpora lutea. Following luteolysis, fresh embryo transfer would require alternative luteal phase support to secure good clinical outcome. Alternatively, good quality embryos obtained after GnRH agonist triggering can be cryopreserved and replaced in following frozen-thawn embryo transfer (FTET) cycles. Thus, also eliminating late onset OHSS due to pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* A female patient who needs IVF to become pregnant.
* Regular menstrual cycle.
* Antral follicular count (AFC) > 18
* Following treatment with follitropin beta more than 18 follicles ≥ 11 mm will develop.

Exclusion Criteria:

* Hypersensitivity to the active substance or to any of the medications used.
* Tumors of the ovary, breast, uterus, pituitary or hypothalamus.
* Pregnancy.
* Abnormal (not menstrual) vaginal bleeding without a known/diagnosed cause.
* Primary ovarian failure.
* Ovarian cysts or enlarged ovaries.
* A history of Ovarian Hyperstimulation Syndrome (OHSS).
* A previous COS cycle that resulted in more than 30 follicles > 11 mm measured by ultrasound examination.
* Fibroid tumours of the uterus incompatible with pregnancy.
* Malformations of the reproductive organs incompatible with pregnancy

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2012-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety: The adverse event is the development of OHSS following oocyte retrieval. | 12 day from GnRH agonist trigger day.
  OHSS usually occurs a few days following oocyte retrieval, and is not a threat once menses start.

SECONDARY OUTCOMES:
Ongoing pregnancies following FTET cycles of cryopreserved embryos obtained following one treatment cycle of follitropin beta. | One month from embryo transfer date

CONTACTS AND LOCATIONS:
Overall Officials: Shahar Kol, MD, Principal Investigator — Elisha Hospital, Haifa, Israel
Locations (1):
- IVF Unit, Elisha Hospital, Haifa, Israel, Israel